CLINICAL TRIAL: NCT03331601
Title: Evaluation of 68GaNOTA-Anti-HER2 VHH1 Uptake in Brain Metastasis of Cancer Patients
Brief Title: Evaluation of 68-GaNOTA-Anti-HER2 VHH1 Uptake in Brain Metastasis of Cancer Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: UZBRU_VHH1_2; 2015-002328-24 (EudraCT Number)
Record Dates: First submitted 2017-10-24; First posted 2017-11-06 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-02

CONDITIONS: Carcinoma; Receptor, ErbB-2
Keywords: Brain metastasis; HER2
MeSH Terms: conditions — Carcinoma; Brain Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: 68GaNOTA-Anti-HER2 VHH1 — Injection of the radiopharmaceutical and PET/CT 90 min post injection

SUMMARY:
This study investigates the uptake of the radiopharmaceutical 68-GaNOTA-Anti-HER2 VHH1 in brain metastasis using PET/CT imaging. Patients with HER2-positive and HER2-negative cancer will be included and the uptake in their lesions will be compared.

Optional 68-GaNOTA-Anti-HER2 VHH1 scans may be performed during or after treatment, at time points 12±6 weeks and 24±9 weeks after the first scan.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have given informed consent
* Age 18 years or older
* Patients with brain metastasized cancer, with at least 1 brain lesion of at least 8 mm maximal diameter, as measured by CT or MRI.
* Patients with potentially HER2-positive cancer. Either a HER2 staining should have been done in standard of care, or sufficient tissue should be available for HER2-staining for study purpose.

Exclusion Criteria:

* Pregnant patients
* Breast feeding patients
* Patients with recent (< 1 week) gastrointestinal disorders with diarrhea as major symptom
* Patients with any serious active infection
* Patients who have any other life-threatening illness or organ system dysfunction, which in the opinion of the investigator would either compromise patient safety or interfere with the evaluation of the test radiopharmaceutical
* Patients who cannot communicate reliably with the investigator
* Patients at increased risk of death from a pre-existing concurrent illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-10-16 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The tumor targeting potential in brain metastasis | 90 min post injection
  The tumor targeting potential in brain metastasis will be visually scored as positive or negative by an experienced nuclear medicine physician, unaware of the HER2-status.
The tumor targeting potential in brain metastasis | 90 min post injection
  The tumor targeting potential in brain metastasis will be assessed quantitatively using Standard Uptake Values (SUV) by an experienced nuclear medicine physician, unaware of the HER2-status.

SECONDARY OUTCOMES:
Change in uptake in brain lesions evaluated by PET/CT scan during or after treatment | up to 2 years after inclusion
  If available, uptake will be evaluated during and after treatment and compared to baseline values. Results will be compared to information of patient's disease course

CONTACTS AND LOCATIONS:
Overall Officials: Tony Lahoutte, MD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- Uz Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Keyaerts M, Xavier C, Heemskerk J, Devoogdt N, Everaert H, Ackaert C, Vanhoeij M, Duhoux FP, Gevaert T, Simon P, Schallier D, Fontaine C, Vaneycken I, Vanhove C, De Greve J, Lamote J, Caveliers V, Lahoutte T. Phase I Study of 68Ga-HER2-Nanobody for PET/CT Assessment of HER2 Expression in Breast Carcinoma. J Nucl Med. 2016 Jan;57(1):27-33. doi: 10.2967/jnumed.115.162024. Epub 2015 Oct 8. PMID 26449837